CLINICAL TRIAL: NCT04023981
Title: Parafricta Bootees Compared to UK Standard Care to Prevent Heel Pressure Ulcers: a Multicentre Pragmatic Randomised Controlled Trial With Blinded Assessment at Three Days and at Fourteen Days.
Brief Title: Parafricta Bootees vs UK Standard Care to Prevent Heel Pressure Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting eligible participants
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Welsh Wound Innovation Centre (Unknown)
Responsible Party: Principal Investigator, Dr Grace Carolan-Rees, Professor Grace Carolan-Rees, Cardiff and Vale University Health Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WA/17/0051
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pressure Ulcer; Pressure Injury; Heel Ulcer
Keywords: Parafricta; Pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment of the primary study outcome was by independent blinded assessment of digital photographic images, by assessors who did not undertake study visits and who were unaware of the participant's allocated treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care alone (No Intervention): Patients randomly allocated to standard care will be cared for on the appropriate mattress indicated for use in that participating centre according to local policy e.g. foam mattress or dynamic air mattress. Standard care may also include a mattress overlay or the use of a wedge or pillows to maintain the position of the participant, or pressure offloading boots on the foot if the need arises during the study period.
- Parafricta bootees plus standard care (Experimental): Patients randomly allocated to Parafricta plus standard care will be cared for on the appropriate mattress as above and care may possibly include a mattress overlay or the use of a wedge or pillows. Participants will in addition be issued with Parafricta bootees (one pair and up to two spare pairs). The patient and clinical staff and the patient's carers will be instructed in the use of Parafricta bootees, which are intended to be worn throughout the day and night and removed only for normal daily washing or examination of the patient's feet. Either the slip-on bootees or the Velco-closure bootees will be selected for the participant at the judgment of the clinical ward nurses.
  Interventions: Device: Parafricta bootees

INTERVENTIONS:
Device: Parafricta bootees — Parafricta bootees are a medical device designed to eliminate skin damage due to friction and shear. The basis of Parafricta bootees is a low friction material and bi-layer construction to make the material of the bootee slide on itself when movement of the foot would otherwise bring friction and shear to bear on the skin.
  Arms: Parafricta bootees plus standard care

SUMMARY:
This randomised study will assess whether Parafricta bootees, when used in addition to normal standard care, can reduce the incidence of heel PUs in patients at very high risk of skin breakdown. The participant group will be hospital inpatients at high risk of PUs (Waterlow score of 20 or more) who are bedbound and do not have existing heel PUs. The participants will be randomised to an intervention arm using Parafricta plus standard care, or a control arm of standard care only. The primary outcome is incidence of heel PUs at day 3. Secondary outcomes are incidence of PUs at day 14, length of stay, severity of PUs, patient acceptability of device, cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria for this study at the time of recruitment were:

* Adult of age 18 years or over
* Admitted to secondary care in an in-patient hospital (with no specified interval from admission to hospital to study recruitment)
* Bedbound or unable to walk independently and requiring assistance to transfer to a chair
* 'Very high' risk group for pressure ulceration (defined by a Waterlow Score of 20 or more)
* No existing heel pressure ulcers of EPUAP/NPUAP/PPPIA Category 1 or above or any other type of wound on the feet.
* Patient was not being treated with pressure offloading boots.
* Patient was not being treated with a heel cast.

Exclusion Criteria:

• Patients with a single or double lower limb amputation were not eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of heel pressure ulcers of EPUAP NPUAP/PPPIA Category 1 or above | Day 3
  Incidence of heel pressure ulcers of EPUAP NPUAP/PPPIA Category 1 or above on Visit 2 (Day 3), assessed by examination of digital images by two independent expert assessors who are blinded to the participants' allocated treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Carolan-Rees, Prof, Study Director — Cedar, Cardiff & Vale University Health Board
Locations (1):
- Cedar, Cardiff & Vale University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided